CLINICAL TRIAL: NCT01484717
Title: Interactive Voice Response Technology to Mobilize Contingency Management for Smoking Cessation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UConn Health (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11-132-2; R21DA029215 (NIH)
Record Dates: First submitted 2011-11-30; First posted 2011-12-02 (Estimated); Last update posted 2017-02-20 (Actual); Status verified 2017-02

CONDITIONS: Cigarette Smoking
MeSH Terms: conditions — Cigarette Smoking | interventions — Tobacco Use Cessation Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Care (Active Comparator): Telephone counseling plus nicotine patch
  Interventions: Drug: transdermal nicotine; Behavioral: Telephone counseling
- Contingency management for abstinence from cigarettes (Experimental): Telephone counseling and nicotine patch plus contingency management
  Interventions: Behavioral: contingency management for smoking abstinence; Drug: transdermal nicotine; Behavioral: Telephone counseling

INTERVENTIONS:
Behavioral: contingency management for smoking abstinence — Participants earn the chance to win prizes for breath samples that test negative for cigarette smoking.
  Arms: Contingency management for abstinence from cigarettes
Drug: transdermal nicotine — Participants receive an 8 week supply of transdermal nicotine [21 mg patches (4 wks), 14 mg (2 wks), 7 mg (2 wks)].
Behavioral: Telephone counseling — Participants receive brief twice weekly telephone counseling.

SUMMARY:
Cigarette smoking remains the most common source of preventable morbidity and mortality in the United States, with in excess of $167 billion in economic costs per year. Contingency management (CM), in which tangible incentives are provided contingent on a target behavior like abstinence, is highly efficacious in improving substance abuse treatment outcomes and is receiving increased attention for smoking cessation. Expired carbon monoxide (CO) is the most common objective smoking status test used in smoking research and treatment. Unfortunately, multiple CO tests/day are typically required to detect all smoking and reinforce sustained abstinence. The resulting logistical and resource limitations greatly limit the application of this potentially powerful quit smoking toolset. This study addresses these limitations by examining the effectiveness of using interactive voice response technology (IVR) to implement CM. Smokers who want to quit (N = 90 randomized) will receive 2 quit preparation sessions based on public health guidelines for smoking cessation and set a target quit date. Participants will be randomly assigned to 1 of 2 treatment conditions: (a) IVR-S consisting of objective smoking status monitoring using IVR, telephone counseling and transdermal nicotine and (b) IVR-CM, consisting of the same monitoring, telephone counseling and transdermal nicotine plus IVR-based CM for smoking abstinence. It is hypothesized that abstinence rates will be higher in the IVR-CM condition compared to the IVR-S, supporting a combined IVR CM approach, and thereby greatly increasing the applicability of these powerful smoking cessation tools.

ELIGIBILITY:
Inclusion Criteria:

* regular cigarette smoker
* age ≥ 18
* mailing address & valid photo I.D.
* want transdermal nicotine

Exclusion Criteria:

* not English speaking
* in recovery for pathological gambling
* contraindication for transdermal nicotine
* female who is pregnant, nursing a child, or not using effective contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2012-01; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Longest duration of abstinence | Week 24

CONTACTS AND LOCATIONS:
Overall Officials: Sheila Alessi, Ph.D., Principal Investigator — UConn Health
Locations (1):
- University of Connecticut Health Center, Farmington, Connecticut, United States

REFERENCES:
- [Derived] Alessi SM, Rash CJ. Treatment Satisfaction in a Randomized Clinical Trial of mHealth Smoking Abstinence Reinforcement. J Subst Abuse Treat. 2017 Jan;72:103-110. doi: 10.1016/j.jsat.2016.06.013. Epub 2016 Jul 4. PMID 27449226